CLINICAL TRIAL: NCT00932958
Title: Physicians International CCTA Utilization Registry
Brief Title: Physicians International Coronary Computed Tomography Angiography (CCTA) Utilization Registry
Acronym: BIGPICTURE
Status: Completed | Type: Observational
Sponsor: MDDX LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: bigPICTURE
Record Dates: First submitted 2009-07-05; First posted 2009-07-07 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All comers >18 yrs old: This study is observational, studying patients who are already scheduled to undergo CCTA. Minors and those unable to consent to the study are excluded.

SUMMARY:
This protocol describes an observational study whose goal is to collect de-identified Coronary CT Angiography (CCTA) acquisition factors and interpretations (findings) from several hundred U.S. and international imaging facilities. The study uses an electronic data capture tool to collect de-identified CCTA utilization parameters and clinical findings in order to create a multi-center registry. This registry will be used for scientific analysis and publication of pertinent medical trends such as CT utilization, radiation dose, and common cardiovascular findings. The registry will be used to determine areas of interest for future randomized controlled trials.

All data will be collected with patient identifiers removed and in complete accordance with HIPAA regulations. All data will be analyzed in aggregate, thus further minimizing the risk of patient confidentiality violations.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants who are able and willing to consent for themselves
* Patients scheduled for CCTA examination

Exclusion Criteria:

* Patients who did not complete the planned CT imaging procedure due to mechanical error of the CT machine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 or older) who are scheduled to undergo a CCTA imaging procedure.
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
CCTA utilization parameters and clinical findings | Two years

SECONDARY OUTCOMES:
90 day MACE, Intended Care Management and Cost Effectiveness for cardiologists interpreting their CCTA studies | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gebow, PhD, Study Director — MDDX LLC
Locations (1):
- MDDX, San Francisco, California, United States